**Title:** Evaluation of pain alleviating strategies during allergy shots (Subcutaneous immunotherapy): A randomized controlled study (**P**ain **P**erception with **A**llergy **S**hot **Techniques**: PPAST)

# **Principal Investigator**

Jennifer Pfieffer MSN, APRN, PCNS-BC, CPEN

# **Co-Investigators**

- Karen Gee BSN, RN, CPN
- Kristine Wehmeier BSN, RN, AE-C
- Emily Hoehn BSN, RN, CPN
- Monarie Lacanilao BSN, RN
- Tracy DeSanto BSN, RN, CPN
- Tara Spruill MSN, RN, CPN
- Jamie Thibodeaux BSN, RN, CPN
- Amanda Davis BSN, RN Ejaz Yousef MD

## **Research Coordinators**

- Isabel Delgado, BSH
- Elizabeth DeLuca, BSN, RN, CCRC
- Mary Warde, BSN, RN, CCRC

# **Project Consultant / Data Analyst**

Keith Fishlock MSN,ARNP,PCNS-BC, FNP-BC

# **Rationale and Purpose**

Subcutaneous Immunotherapy (allergy injections) is a potentially disease-modifying therapy that is effective for the treatment of allergic rhinitis/conjunctivitis, allergic asthma and stinging insect hypersensitivity. Pain, which results from the irritation of nearby nerves is a common concern of patients, particularly in children, during or after the injections. This can be a stressful and negative experience for the children. There are various techniques available to minimize pain in general. However, there is a lack of published research on how to use these techniques in children receiving allergy injections. The purpose of this study is to evaluate and compare the efficacy of the standard of care method (Ethyl Chloride/Pain Ease Spray) and three non-pharmacological pain control devices (Buzzy Bee I, Buzzy Bee II and Shot Blocker) in decreasing the perception of pain during subcutaneous allergy injection in a pediatric allergy/immunology clinic setting.

#### **Objective**

 Evaluate and compare the effectiveness of utilizing various techniques to reduce the perception of pain during subcutaneous allergy injections in children

# **Possible Risks and Benefits**

Risk Assessment

The risks associated with study participation are consistent with standard of care risks.
 Potential risk for the study participants may be possible allergic reaction/skin irritation from the cold spray or ice pack or an increased level of anxiety.

#### Benefits Assessment

The potential benefit associated with this research study includes a better understanding
of study participant's response to their assigned distraction technique. This study may
help identify which technique is more beneficial to use in children receiving
subcutaneous immunotherapy to decrease the perception of pain and reduce anxiety
related to immunotherapy treatment.

# **Study Design and Duration**

This is a randomized controlled study. Approximately 100 children, age 4 – 17 years, who are currently receiving subcutaneous immunotherapy, will randomly select a blinded envelope which assigns the distraction technique to be utilized during their study participation. There will be 25 envelopes assigned to each study group for a total of 100 envelopes. Each envelope will contain a paper with a colored sticker for the associated group assignment and number sequence.

The distribution of group assignment by number sequence and color is as follows:

- Interventional Groups
  - 1. Shot Blocker® # 1-25 (RED)
  - 2. Buzzy I (vibrating only) # 26-50 (GREEN)
  - 3. Buzzy II (vibrating and ice wings) #51-75 (BLUE)
- Control Group
  - 4. Ethyl Chloride/Pain Ease Spray # 76-100 (YELLOW)

The three interventional groups are currently marketed distraction devices. The control group is the current clinical standard of care option for pre-allergy injection application.

The study consists of two visits. Both visits will be conducted during the participants routine clinic visit for allergy injections. At the first visit the investigator will assess eligibility. An overview of the study requirements will be provided to parent/child and consent/assent will be obtained.

During the second visit, the child will be randomized to a distraction technique or standard of care group to be utilized with the allergy injection(s) administered at this visit. Adherence with institutional allergy injection guidelines will be maintained. Prior to the application of the distraction method, the investigator will interview the parent to collect data related to demographic information and their child's current allergy health and treatment regime. The child's pain perception will be assessed before and after the allergy injection. The parent's perception of their child's pain will be assessed after the allergy injection. The investigator will provide information on the application of the randomized method and will provide instruction on the completion of the pain scales and questionnaires. The investigator and study staff will not indicate a method preference or guide the child or parent with their pain level responses. After completion of the second visit, the child's study participation is complete.

# **Inclusion & Exclusion Criteria**

**Inclusion Criteria** 

- Children aged 4-17 years on injection immunotherapy
- A minimum of three allergy injection injections prior to enrollment at Visit 1

• Child accompanied by parent or legal guardian

#### **Exclusion Criteria**

- Children with a known pain or sensory disorders
- · Developmental delays lacking necessary cognitive ability
- Administration of any form of pain analgesic within eight hours of randomization at Visit 2

# **Study Procedures**

### Visit 1:

Children aged 4-17 years who present to receive their injection(s) in the allergy clinic will be screened by the Principal Investigator or Co-Investigator for study inclusion and exclusion criteria. During their routine post-allergy injection 30-minute wait time, the investigator and the research coordinator will provide the parent and child with an overview of the study design, the risk and benefits assessment and study requirements. The investigator will advise the parent/child of the pain analgesic administration exclusion for the randomization visit. After obtaining parental permission and child assent, the child will be considered enrolled in the study. A subject ID will be assigned. A visible mark placed on the child's allergy injection chart will indicate the child is ready to be randomized at their next routine allergy injection visit.

#### Visit 2:

At a future allergy injection clinic visit the parent and the child will be asked if the child took any pain-relieving medicines, like Tylenol or Advil, within eight hours before coming to the clinic. If the participant needed this kind of medicine, the allergy shot appointment will be the same as before the study.

Study visit 2 will be completed at another routine allergy shot appointment. Preferably the next scheduled allergy injection visit.

If the participant did **not** take any pain relieving medicine within the previous eight hours, visit 2 will continue. The participants study group assignment will be determined. The envelopes identifying the four group assignments will be coded by number and color. The child will be presented with a basket containing all the envelopes. The investigator will instruct the child to select one envelope from the basket. The envelope selected at random by the child will determine the distraction method to be utilized prior to the allergy injection(s). The possible group assignments, one of three currently marketed distraction devices or the control group utilizing the current standard of care option, are listed below and are further detailed in Attachments I – III.

The four study groups are:

- > Interventional Groups
  - 1. Shot Blocker®
  - 2. Buzzy I (with ice pack-wings)
  - 3. Buzzy II (without ice pack-wings)
- Control Group
  - 4. Ethyl Chloride/Pain Ease Spray

# Before applying the assigned distraction method:

- Prior to randomization, the investigator will interview the parent to obtain the information needed to complete the Parent Demographic-Health-Treatment Questionnaire (Attachment V). The investigator will review the responses for any indicator of study ineligibility, ie, analgesic medication window.
- The investigator or study staff will review the Wong-Baker FACES Pain Rating Scale with the child. The child will be given a Wong-Baker FACES Pain Rating Scale form and asked to circle the face which most closely matches their current level of pain awareness prior to any intervention. (Attachment IV-a)
- The investigator or study staff will review the Numeric Pain Rating Scale (Attachment IV-b) with the parent. The parent will be instructed to circle the number on the scale which most closely matches their perception of their child's pain level immediately after receiving the allergy injection.

# Application of the distraction method and administration of the allergy injection:

- The investigator will apply the assigned distraction method per method specifications to the injection site area (subcutaneous region of the back of the upper arm).
- The investigator will administer the subcutaneous allergy injection(s) within the time frame specified for the assigned distraction device utilized or per the standard of care guidelines for the Pain Ease Spray, as appropriate. If the child's treatment plan includes more than one injection, the assigned group technique will be utilized for all injections at the visit.

# Post allergy injection procedures:

- Immediately following the allergy injection, the child will be provided with a second Wong-Baker FACES Pain Rating Scale form and be asked to circle the face which most closely matches their post-injection level of pain awareness.
- Immediately following the allergy injection, the parent will be reminded to circle the number on the Numeric Pain Rating Scale which most closely matches their perception of the child's post-injection pain level.
- The participant and parent will then complete the routine 30 minute wait time for post allergy injections.

Study participation is complete at the end of Visit 2.

# **Prohibited Medications**

Analgesic medications administered within eight hours of Visit 2 are prohibited.

# Adverse Event (AE)

An AE is any unfavorable and unintended sign, symptom temporally associated with the use of the study technique and does not imply judgment about causality.

AE's associated with the randomized intervention will be collected at Visit 2. The AE's relationship to the distraction technique will be assessed using the following guidelines for causality and grading severity. AE's related to the allergy injection will not be captured in this study.

**AE Relationship to Study Distraction Technique Guide** 

| Relationship to Study Distraction Technique | Comment |
|---|---|
| Definitely | An event that follows a reasonable temporal sequence from administration of the study distraction technique; that follows a known or expected response pattern to the suspected study distraction technique; that is confirmed by stopping the use of the study distraction technique; and this is not explained by any other reasonable hypothesis. |
| Probably | An event that follows a reasonable temporal sequence from administration of the study distraction technique; that follows a known or expected response pattern to the suspected study technique; that is confirmed by stopping the use of the study distraction technique; and that is unlikely to be explained by the known characteristics of the subject's clinical state or by other interventions. |
| Possibly | An event that follows a reasonable temporal sequence from administration of the study distraction technique; that follows a known or expected response pattern to that suspected study distraction technique.; but that could readily have been produced by a number of other factors. |
| Unrelated | An event that can be determined with certainty to have no relationship to the study distraction technique. |

**AE Severity Grading** 

| Severity (Toxicity Grade) | Description |
|---|---|
| Mild (1) | Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated |
| Moderate (2) | Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate Instrumental activities of daily living (e.g., preparing meals, using the telephone, managing money) |
| Severe (3) | Severe or medically significant but not immediately life threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care activities of daily living (e.g., bathing, dressing, feeding self, using toilet, taking medications) |

# <u>Discontinuation and Replacement of study participants</u>

A child has the right to withdraw from study participation prior to the completion of Visit 2. Early withdrawal participants will be replaced one to one.

# Participant ID assignment

The study participants will receive a Participant ID at Visit 1 which will be used for all data collection. The Participant ID used will range from 001 to 100. If a study participant withdraws before the completion of Visit 2, the Participant and associated group assignment will be replaced. Replacement Participant ID's will be sequential beginning with the number 101.

# **Data Collection**

Medication administration data collected will be limited to the participant's current immunotherapy vial and dosing, distraction method utilized, site of the application method and, if applicable, antihistamine use and pain medication use. Demographic data collected will be age, race and gender. Symptom and health data point collection will target allergy injection reactions and the presence of allergic rhinitis, asthma and atopic dermatitis. (Refer to Attachment V). Pain perception data will be collected from both the child and parent using facial and numeric pain scales (Refer to Attachment IV).

All data collected will be entered into an EXCEL data collection tool and stored on password protected, secure computers. The data will accessible only to the investigators and research coordinators in the study.

### **Data Analysis**

Quantitative component data collected and evaluated for this study will include the number of patient participants within the allergy department, randomized interventions used, diagnoses including allergic rhinitis, asthma and atopic dermatitis, immunotherapy medication and dose, antihistamine and pain medication utilization, patient and parental pain scores, adverse reactions, age, race, and gender.

Quantitative component data collected for this study will be extracted into Microsoft Excel spreadsheets and analyzed using Excel functions. Target population demographic characteristics will be analyzed using descriptive statistics by the principal investigator with the level of significance set at <0.05.

All information collected as part of evaluating the impact of this study will be aggregated data from the project participants and will not include any potential patient identifiers. Participant confidentiality will be assured by coding the participants using individual identification numbers for any analysis activities occurring outside of the electronic health record. This information will be stored in accordance with Nemours IRB policies and procedures. The Excel files containing codified data without protected health information (PHI) will be stored in password protected files at Nemours, on a password protected desktop computer in a locked office space accessible only by the principal investigator and study designees. The risk to patients participating in this project will be no different from the risks of patients receiving standard care.

# **Informed Consent Process**

- Children who meet study criteria will be identified by Principal Investigator or Co-Investigator in the allergy clinic.
- Parents/guardians and child will be given an overview of the study, participation requirements, and complete information on being a voluntary participant in a research study. They will be given an opportunity to read the consent form, have questions answered and decide if they want their child to participate.
- If both the parent and child are interested in participating in the study, one parent/legal guardian will be asked to sign a Parental Permission and Consent Form.
- Children between the ages of 7 and 17 who verbalize understanding and are agreeable to the Assent information and study expectations will be asked to sign a Child Assent or Adolescent Assent Form.
- The Principal Investigator, Co-Investigator or Research Coordinator obtaining consent will witness the parent and child signatures, will sign both documents and provide copies of the signed consent/assent to the parent and child.

# **Participating Sites**

The study will be conducted at Nemours Children's Specialty Care in the pediatric allergy clinics locations:

- Jacksonville Downtown
- Jacksonville South
- Fleming Island

### **Literature Cited**

Angela Li, Zorash Montaño, Vincent J Chen, and Jeffrey I Gold: Virtual reality and pain management: current trends and future Directions:; Pain Manag. 2011 March; 1(2): 147–157

Rasha Srouji, Savithiri Ratnapalan, and Suzan Schneeweiss: Pain in Children: Assessment and Nonpharmacological Management.. International Journal of Pediatrics; Volume 2010

Psychological interventions for needle-related procedural pain and distress in children and adolescents:Cochrane Systematic Review - Intervention Version published: 04 October 2018

<u>Ariane Ballard</u>,<sup>2</sup> <u>Christelle Khadra</u>, <u>Samara Adler</u>, <u>Evelyne Doyon-Trottier</u>, and <u>Sylvie Le May</u>:Efficacy of the Buzzy® device for pain management of children during needle-related procedures: a systematic review protocol; <u>Syst Rev</u>. 2018; 7: 78.

Shomaker K, Dutton S, Mark M. Pain prevalence and treatment patterns in a US children's hospital. Hosp Pediatr 2015;5:363–7.

Stevens BJ, Yamada J, Estabrooks CA, Stinson J, Campbell F, Scott SD, Cummings G; CIHR Team in Children's Pain. Pain in hospitalized children: effect of a multidimensional knowledge translation strategy on pain process and clinical outcomes. PAIN 2014;155:60–8.

Vessey JA, Carlson KL, McGill J. Use of distraction with children during an acute pain experience. *Nursing Research*. 1994;43(6):369–372

Cohen LL, Blount RL, Cohen RJ, Schaen ER, Zaff JF. Comparative study of distraction versus topical anesthesia for pediatric pain management during immunizations. *Health Psychology*. 1999;18(6):591–598.

# **Attachments**:

### ShotBlocker®

ShotBlocker instantly reduces needle pain and anxiety associated with injections.

ShotBlocker distracts and comforts patients of all ages receiving intramuscular or subcutaneous injections to lessen the perceived pain and anxiety. ShotBlocker is an innovative, patented device that is both simple and easy-to-use.

#### Features and Benefits

- Simple Design One ShotBlocker per patient is all you need.
- Easy to Use Just press ShotBlocker firmly over the injection site and give the injection through or near the opening.
- Immediate Effect The contact points on the underside create an immediate distracting effect. No waiting for topical anesthetics to take effect.
- Versatility Useful in intramuscular injections, subcutaneous injections and other procedures that include a painful needle poke.
- Cost Benefit Less costly than anesthetic creams or freezing sprays. (Faster, too.)
- Smiles On Your Patient's Faces Invented by a pediatrician to lessen the pain and anxiety experienced by his patients.
- It Really Works!

# **Product Offering**

**#8050** - Box of 50 **#8100** - Box of 100







Phone 1.800.551.6810

Fax 1.800.455.5678

Web www.BionixMed.com

### How ShotBlocker® Works

ShotBlocker is a novel application of the gate control theory of pain management. ShotBlocker is a flexible plastic disk that has a number of blunt contact points on its underside. When pressed firmly against the patient's skin at the injection site, ShotBlocker saturates the sensory signals distracting the patient from the pain signals caused by the needle poke.



### How to Use





- 1. Select the injection site and prep the skin as usual.
- 2. Hold ShotBlocker so that the blunt contact points touch the patient's skin at the injection site.
- 3. Press ShotBlocker FIRMLY against the skin. (A)

  DO NOT MOVE OR REMOVE SHOTBLOCKER UNTIL
  THE INJECTION HAS BEEN COMPLETED.
- 4. Immediately administer the injection in the usual manner through or near the central opening of ShotBlocker. For subcutaneous injections, angle the needle as needed to give the injection. (B)
  - IF MORE THAN 20 SECONDS ELAPSE BETWEEN THE PLACEMENT OF SHOTBLOCKER AND THE INJECTION, COMPLETELY REMOVE SHOTBLOCKER FROM THE SKIN. REPEAT THE PROCESS BEGINNING WITH STEP 2.
- After you have completed the injection and withdrawn the needle, remove and discard ShotBlocker.





II – Buzzy Bee I (with ice pack-wings) and Buzzy Bee II (without ice pack-wings)







Developed by a physician, Buzzy® is a reusable device for minor aches and pains.

tended to be used by a single user.

Bring with you to the doctor; or use at home for:

- # STINGS
- SPLINTERS

#### BuzzyHelps.com

Home Use Rev. 02.01.17

Wings will stay frozen 10 minutes at room temperature. For best pain relief, the Wings must be frozen solid to avoid absorbing vibration.

Face the blue or smooth side of the Wings toward the skin for more rumbing power. If sensitive to cold, the soft side of the wings should face the skin.

Tip: For long procedures or for medications that burn or sting, prepare additional Wings.

Store folded Wings in freezer. Gel inside Wings is a non-taxic, safe, food-grade product that may deteriorate if not stored properly.

Note: To transport, place the Wings between the ColdToGo bag blue toe inserts (sold separately), or between 2 commercial cold packs (sold separately) to maintain frazen temperature.

Our Comfort Strate:

Our Comfort Strap is a revisable, single-handed tourniquet, smooth and pirich free. To use, 1. Loop the Comfort Stop around the crm, passing one end finough the slit in the other. 2. Hold the slit and pull the other end through until the desired tension is reached, then releases the slitted end. 3. To lock the Comfort Strop in position, releases the tension from the long end. 4. To release, simply pull gently on the short end and the Comfort Strop will fall gway.

INDICATIONS FOR USE ......CONTRAINDICATIONS, WARNINGS, AND CAUTIONS ...
ICE WINGS .......
COMFORT STRAP.... DIRECTIONS FOR USE .. BUZZY PLACEMENT ..... SHOTS ... STOMACH INJECTIONS ... FOR ACHES AND PAINS ..... FINGER STICKS, SPLINTERS . BURNING, ITCHING TROUBLESHOOTING. ORDERING, GUARANTEE .



#### DIRECTIONS FOR USE:



Immediately before use, remove the Immediately before use, remove the Wings from the freezer and attach behind Buzzy® on the hook. Activate by firmly pressing button on top of Buzzy®. Press a second time to turn, Buzzy® off.

Buzzy® has an energy saving outomatic shut-off after 3 minutes of press the button on top of Buzzy® to

reconce vibration.

Buzzy comes with a sticone Comfort Stop to hold Buzzy in place on extentiliss 1, toop the Comfort Stop pround the arm, passing one end through the sit in the other. 2, Hold the sit and pull the other end through until the desired tension is a roched, their release the stitled end. 3, To lock the Comfort Stop in position, release the tension is not the large end. 4. To release, simply pull gently on the short end and the Comfort Stop will fall awary.

Use Buzzy® only on clean, unbroken skin. The stripes on Buzzy®, or bottom end should be closest to the procedure, and the head on Buzzy® and switch farthest away. Tip: For best results, center the bigger rounded end of Buzzy® directly next to

#### INDICATIONS FOR USE:

INVICATIONS PUR USE:
Controls pain associated with injections |venipuncture, IV starts, cosmetic procedures| and the temporary relief of minor injuries [missile or tendon aches, splinters and bee strings]. Also intended to toor impolarisal poin caused by trigger points, restricted motion and musicle tension.

Fold Wings and STORE IN FREEZER. Wings must be frozen sold for best effect. Personal Buzzy<sup>®</sup> units coms with universal personal loe Wings & Comfort Strap.

WARNINGS: For intended use only • Direct or prolonged application of ice could vasoconstrict or alter lab values.

CONTRAINDICATIONS: Do not use in the presence of unexplained calf pain. Consult a physician. • This device should not be used over swollen or inflamed areas or skin eruptions. • Do not place directly on a thermal burn • Do not use ice pack with underlying sensitivities to ice or cold (e.g. Sickle Cell Disease, Raynaud's Disease).

CAUTIONS: Store in a cool, dry place.

### Buzzy PLACEMENT:







The Buzzv® The Buzzy® physiologic blockade works best when placed "between the brain and the pain" in the same nerve area as the pain. On arms and shoulders, nerves run from fingers to shoulders to the spine. For the chest and back, the nerves run from the center of the chest or stomach horizontally to the back. On the thighs, the nerves run diagonally from the inner thigh around to the back to the spine.

For children: For best results, let children hold Buzzy® in advance for familiarity, and let them choose whether or not to use the ice pack.

For shots: Switch on to activate the vibration, and then place Buzzy® on the site of the shot. Leave for 15 seconds for surface shots - 60 seconds for deeper injections. Immediately before cleaning the site, move Buzzy® proximal (closer to the head) to the pain location, and press in place throughout cleaning and getting the shot.





For children who get their shots sitting up, a parent can put an arm around the shoulders to hold Buzzy® For injections in the stomach: [ Place Buzzy® lateral to the shot (i.e., belly button, the shot, and then Buzzy®



#### For Aches and Pains:

Apply directly to sore muscles for maximum of 10 minutes. Hold in place or attach with strap. Buzzy® has an energy saving automatic shut-off after 3 minutes of constant use. Simply press the button on top of Buzzy® to reactivate vibration.

For additional placement information, please visit: bzy.fyi/howto

For finger sticks or splinter removal: Switch on to activate the vibration, and then press Buzzy® on the palm with the bottom end toward the finger. Leave in place throughout deaning and doing the procedure.



7

For burning or itching: Like any cold and warm therapy application, Buzzy® can be helpful for burning or itching. For insect bites or medications that cause burning or itching, take frazen Wings and massage the vibrating Buzzy<sup>®</sup>/Wings combination directly on the site. Rub or press in place until the area feels better. Do not place Buzzy® directly on a thermal burn.



#### For IVs or phlebotomy:

Switch on to activate the vibration, and then place Buzzy<sup>10</sup> proximal (above) to the pain location. Press in place or tuck under tourniquet before immediately cleaning and obtaining access. Pass any tourniquet through slot to secure Buzzy® to arm. Do not [ put directly on site of access.



Buzzy® is a personal consumer product intended to be used by a single user. Buzzy® may be cleaned with alcohol based sanitation wipes. Do not autoclave. Do not immerse in liquid. Sailed wings should be disposed of and replaced.

#### BATTERIES:

Buzzy's batteries will last at full strength about 20 hours. For best pain relief, replace batteries when vibration weakens. Unscrew the back using a Phillips head screwdriver to remove back panel. Buzzy® is powered by 2 alkaline AAA batteries. Remove batteries if Buzzy is not being used for extended period of time.

If you are having trouble powering on your Buzzy® unit, please open up your Buzzy®, remove the batteries, bend the battery tabs inward, and replace the batteries.

**TROUBLESHOOTING:**When used with care, Buzzy® should last years. If Buzzy® is dropped repeatedly, howevers, the metal that holds the batteries in place can bend. If Buzzy® falls to function after a fall, try prinching bottery clip in to restore contact.

HOW TO ORDER /ADDITIONAL INFORMATION: Please visit our website BuzzyHelps.com for a comple FAQ's, other pain management tips, how-to videos, accessories, replacement parts, and more!

GUARANTEE:
Previous medical history and initiasic physiologic differences may make Rizzy® less effective for some people. If not completely satisfied, return within finese months to place of parchase for a full refund, or contact us of the address below.

MMJ Labs 195 Arizona Ave NE, LW 08 Atlanta, GA 30307, U.S.A. BuzzyHelps.com info@mmilabs.com 877.805.2899

US Patented British Patent No. 2455695 RM-1910, 1248064500200, 1248064500100 Arthotzed European Representative MPC INTERNATIONAL S.A.

26, Bovlevard Reyal 52449 (L025/48URG Tel. +252 22 99 99 5546 | www

reposes Type B Applied Part

8.

# III – Ethyl chloride spray





Rx only Invert the bottle while spraying.

# INDICATIONS FOR USE:

INDICATIONS FOR USE:
Gabauer's Ethyl Chloride is a vapiocolant (skin
retrigerart) intended for topical application to control
pain associated with injections, starting IV's and
venipuncture, minor surgical procedures (such as
lancing bolls, or incision and drainage of small
absessess), and the temporary relief of minor sports
injurios. It is also intended for use as a counterinitant is
the management of mydiascial pain, restricted motion
and muscle tension.

# PRECAUTIONS:

PRECAUTIONS:
Do not sprey in eyes. Inhalation of eithyl chloride should be avoiled as it may produce natrodic and general anesthetic effects, and may produce deep anesthesia or fatal coma with respiratory or cardiac arrest. Ethyl chloride is FLAMMABLE and should never be used in the presence of an open fiame or electrical cautery equipment. When used to produce local freezing of tissues, adjacent skin areas should be protected by an application of petrolarum. The thawing process may be paintful, and freezing may lower local resistance to infection and delay healing.

#### ADVERSE REACTIONS:

Cutaneous sensitization may occur but appears to be extremely rare. Freezing can occasionally after skin pigmentation.

CONTRAINDICATIONS: Ethyl Chloride is contraindicated history of hypersensitivity to it. . Ited in individuals with a

#### WARNINGS:

WARNINGS:
For external use only. Do not spray in the eyes. Skin absorption of eithyl chioride can occur; no cases of chronic potsoning have been reported. Eithyl chioride is known as a liver and kidney toxin; long-term exposure may cause liver or kidney damage.

WARNING: This product contains a chemical known to the State of California to cause cancer.

KEEP OUT OF THE REACH OF CHILDREN

### DIRECTIONS FOR USE:

To apply Gebauer's Ethyl Chloride from a bottle, hold the bottle bottle, hold the bottle inverted while spraying. Open the dispenseal spring valve completely altowing the Ethyl Chloride to flow from the bottle.



1. PRE-INJECTION ANESTHESIA Prepare the syringe. Swab the treatment area with

Continued\*

(2)

an ansieptic. Spray the treatment area with Gebauer's Ethyl Chloride continuously for 3 to 7 seconds from a distance of 3 to 9 inches (8 to 23 cm). Spray the area until the skin just turns white; do not trost the skin and quickly introduce the needle with the skin taut. The directions are also to be followed for other types of needle insertion procedures such as starting IV's and venipuncture. TOPICAL ANESTHESIA IN MINOR SURGERY:

TOPICAL ANESTHESIA IN MINOR SURGERY: Clean the operative sits with a suitable enriseptic. Apply petrolatum to protect the adjacent area. Spray Gebauer's Elbly (Chloride on the target area continuously for 3 to 7 seconds from a distance of 3 to 9 inches (8 to 25 cm). Spray until the skin just begins to turn white; do not frost the skin and promptly make incision. The ensethetic societo of Babauer's Ethyl Chloride lasts a few seconds to a min it.

TEMPORARY RELIEF OF MINOR SPORTS INJURIES:
The pain of bruises, confusions, swelling and minor sprains may be controlled with Gebauer's Ethyl Choide. The amount of cooling depends on the Josage. Dosage varies with duration of application. The smallest dose needed to produce the desired shed be used. The arreshable effect of withyl střect should be usecí. The anesthetic effect of ethy hilodide rarely lasts more than a few seconds o a minute. This time interval is usually sufficient to help ecuce or releve the initial trauma of the injury. Datermine the extent of the injury (fracture, sprain, sprain, sprain and second of the injury (sprain of 1) to \$100 t

vould loa.

SPRAY AND STRETCH TECHNIQUE FOR

dYOFASCIAL FAIN:

Bobasier's Ethyl Chloride may be used as a
rounteriritant in the management of myotiscial pain,
estricted motion and muscle tension. Clinical
ponditions that may respond to debauer's Ethylades)
could estimate the management of myotiscial pain,
estricted motion and muscle tension. Clinical
ponditions that may respond to debauer's Ethylades)
could estimate the management of the students
coulder, tight hamatrings, sprained anke, tight
nesseler muscles and referred pains due to irritated
rigger points. Relief of pain facilitates early
nobilization and restoration of muscle function.
he Spray and Stretching Chinquia is a therapeutic
ystem that involves three stages: Evaluation,
ignaying and Stretching. The therapeutic value of
as Spray and Stretching Chinquian is a more refective
when the practioner has mastered all of the stages
and explice them in the proper sequence.

Spraying
 Have the patient assume a comfortable position.
 Take precautions to cover the patient's eyes, nose nd mouth if spraying near the face.

Continued.

(3)

(3)

3) Hold the bottle inverted. From a distance of approximately 12 to 18 inches (30 to 45 cm), ain the stream of it meets the skin at an acute angle, lessening the shock of impact.

4) Direct the spray in parallel sweeps 0.5 to 1 inch (1.5 to 2 cm) apara 1 the rate of approximately 4 inches/second/(10 cm/second). Continue until the entire muscle has been covered. The number of sweeps is determined by the size of the muscle three syres yeards be spenially from the muscle attachment over the trigger point, through and over the reference zone.

Passively stretch the muscle during spray application. Gradually increase the force with successive sweeps. As the muscle rotizes, amountly lake up the slack by establishing a new stretch length. It is necessary to reach the full informal length of the muscle is one-pletely inactivate the trigger point and relieve the pâx, apply mosts the procedure. Apply most the procedure. Apply most reatment. For lasting benefit, eliminate any factors that perpetuale the trigger mechanism.

ONTENTS: Ethyl Chloride



CONTENTS: Ethyl Chloride

### STORAGE:

Contents under pressure. Store in a cool place. Do not store above 120°F (50°C). Do not use near fire or flam: or place on hot surfaces. Do not store on or near high frequency ultrasound equipment.

DISPOSAL:
Dispose of in accordance with local, state and nationa regulations.

CAUTION: Federal law restricts this device to sale by or on the ord-



For more information about this product contact Gebauer Company.

Manufactured by:



Cleveland, Ohio 44128 1-800-321-9348 www.gebauer.com ©2014 Gebauer Company REV 01/14

# IV – Data Collection Instruments for pain rating scales – (a) facial (b) numeric





# V – Parent Questionnaire: Demographic – Health – Treatment Questionnaire

| • | nent Worksheet – <i>Attachment V</i><br>MSN, APRN, PCNS-BC, CPEN |
|---|---|
| Participant ID: | Visit 2:/ |
| <u>Demographic – Health – Treatm</u> | nent Questionnaire: Parent Interview |
| _ | parent to complete this questionnaire.<br>ed prior to administering allergy shot. |
| 1. How old is your child? | |
| What race / ethnicity is your child? | |
| What gender is your child? | |
| 4. How long has your child been on allergy shots? (Estimate | e in weeks, months or years) |
| 5. What is the number of allergy shots your child will receiv | ve today? |
| 6. What color vial is your child on? | |
| 7. What is your child's dose for the allergy shot? | |
| 8. What kind of allergy shot is your child receiving – venom | / fire ant / environment? |
| 9. Has your child ever had symptoms after receiving allergy | shots? |
| If yes, explain: | |
| 10. Has your child taken any medication for pain today? | |
| If yes: What was the name and dose of the pain medic | ation? |
| For what reason was the medication given? | |
| What time was the medication given? | |
| 11. Does your child use antihistamine medications? | |
| If yes: What was the name and dose of this medication | n? |
| How often is the medication given? | |
| What time was the medication given? | |
| 11. Please check the 🗌 if your child has any of the following | ng symptoms: |
| ☐ Allergic Rhinitis ☐ Asthma | ☐ Atopic Dermatitis |
| Investigator Signature | Time form completed Date form completed |